CLINICAL TRIAL: NCT05085080
Title: Chinese Neonatal Extracorporeal Life Support Registry (Chi-NELS)
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Chinese Neonatal Network (Other)
Responsible Party: Sponsor
Other Study IDs: Chi-NELS
Record Dates: First submitted 2021-09-06; First posted 2021-10-20 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Extracorporeal Life Support; Neonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extracorporeal life support (ECLS), also known as extracorporeal membrane oxygenation (ECMO), is an extracorporeal technique which provides respiratory and cardiac support to patients with respiratory and/or heart failure. Neonates account for a significant proportion of patients requiring ECLS support. While with unique pathophysiology among newborn infants, neonatal ECLS treatment faces different challenges (such as specific indications, anticoagulation, hemodynamic management, high incidences of complications, ect.) from those of elder children or adults. Though neonatal ECMO has been used in developed countries since 1970s, the introduction of neonatal ECMO in China was not reported until 2010s. While on the other hand, there has been a rapid increase of neonatal ECLS cases and centers in China in the past decade with a huge variation of numbers of cases and quality among different centers. Therefore, there is an urgent need to monitor the use and quality of neonatal ECLS in China. The goal of the Chinese Neonatal Extracorporeal Life Support Registry (Chi-NELS) is to maintain a registry of use of ECLS in active neonatal ECLS centers across China, to support quality improvement of neonatal ELCS, clinical research and regulatory agencies.

DETAILED DESCRIPTION:
This study aims to establish a neonatal ECLS network of all active ECLS centers in China to facilitate standardization of care and collaborative research. On the basis of the network, this prospective comprehensive registry will enroll all neonates who receive ECLS support in participating centers. The indications, managements, complications and outcomes of neonatal ECLS in China will be described in detail, to monitor the development of neonatal ECLS in China, to identify targets for quality improvement, to assist in reducing mortality and morbidity of neonates requiring ECLS support, and to facilitate innovative clinical researches.

ELIGIBILITY:
Inclusion Criteria:

* ≤28 days of life
* receive ECLS support

Exclusion Criteria:

* none

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonate recieved ECLS support
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | From admission to discharge or death, an average of 3 months
  Mortality during NICU

SECONDARY OUTCOMES:
Rate of successful weaning from ECLS | From admission to discharge or dealth, an average of 3 months
  Proportion of infants who were successfully weaning from ECLS
Incidence of mechanical complications | During ECLS, an average of 3 months
  Complication related to the ECLS circuit
Incidence of hemorrhage | From admission to discharge or dealth, an average of 3 months
  Hemorrhage complication including bleeding at gastrointestinal tract, cannulation site, or surgical site
Incidence of brain death | From admission to discharge or dealth, an average of 3 months
  Brain death is diagnosed according to the definition published on critical care medcine in 2011
Incidence of seizure | From admission to discharge or dealth, an average of 3 months
  Seizure was confirmed by EEG
Incidence of diffuse ischemia of central nervous system (CNS) | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with diffuse ischemia of central nervous system (CNS)
Incidence of CNS infarction | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with CNS infarction
Incidence of intraventricular hemorrhage | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with intraventricular hemorrhage
Incidence of renal failure | From admission to discharge or dealth, an average of 3 months
  Proportion of infants renal failure
Incidence of CPR required | From admission to discharge or dealth, an average of 3 months
  Proportion of infants required CPR
Incidence of cardiac arrhythmia | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with cardiac arrhythmia
Incidence of pneumothorax | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with pneumothorax
Incidence of pulmonary hemorrhage | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with pulmonary hemorrhage
Incidence of hemolysis | From admission to discharge or dealth, an average of 3 months
  Proportion of infants with hemolysis
Incidence of limb ischemia | From admission to discharge or dealth, an average of 3 months
  Proportion of infants limb ischemia
Incidence of infection | From admission to discharge or dealth, an average of 3 months
  Infection include pneumonia, sepsis, urinary tract infection, central nervous system infection etc..
Length of hospital stay | From admission to discharge or dealth, an average of 3 months
  Days of hospitalization
Cost of hospital stay | From admission to discharge or dealth, an average of 3 months
  All costs during hospitallization
Length of mechanical ventilation | From admission to discharge or dealth, an average of 3 months
  Days of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Yun Cao, Principal Investigator — Children's Hospital of Fudan University, Shanghai, China